CLINICAL TRIAL: NCT03137615
Title: An Observational Study of the Cardiovascular Response to Infiltration of Local Anaesthetic Into the Nasal Septum in Patients Undergoing Trans-sphenoidal Resection of a Pituitary Lesion
Brief Title: The Cardiovascular Changes Associated With Septal Local Anaesthesia
Status: Completed | Type: Observational
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: STH17059
Record Dates: First submitted 2015-11-20; First posted 2017-05-03 (Actual); Last update posted 2017-05-03 (Actual); Status verified 2017-04

CONDITIONS: Hypothalamic Neoplasms; Pituitary Diseases; Anesthesia, Local
MeSH Terms: conditions — Hypothalamic Neoplasms; Pituitary Diseases | interventions — Anesthesia, Local

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pituitary Surgery: Patients having pituitary gland surgery
  Inclusion criteria - Any adult patient undergoing trans-sphenoidal pituitary surgery.
  Exclusion criteria - Under 16 years of age, pregnancy, uncontrolled hypertension, allergy to any local anaesthetic, patient refusal or revision pituitary surgery
  Interventions: Procedure: Pituitary surgery; Drug: local anaesthetic injection

INTERVENTIONS:
Procedure: Pituitary surgery — Trans-sphenoidal resection of a pituitary gland lesion.
Drug: local anaesthetic injection — The surgeon infiltrates the nasal septum with local anaesthesia as per usual practice. This consists of Moffet's solution and lidocaine with adrenaline (1:200,000).

SUMMARY:
The purpose of this study is to determine the effects on the heart of injecting local anaesthetic into the nose prior to surgery on the pituitary gland?

DETAILED DESCRIPTION:
People sometimes require surgery on their pituitary gland. This is a gland at the base of your brain which secretes hormones. At the Royal Hallamshire Hospital the investigators are currently conducting a study into the effects of local anaesthetic (a medicine which causes numbness) injection on patients undergoing this particular type of operation.

After patients are anaesthetised (asleep) but before surgery starts the surgeon injecst a local anaesthetic solution into the nose. This is routine practice and is done to provide pain relief afterwards and also to decrease the amount of bleeding during the operation to ensure that the surgeon has a good view.

The investigators have known for a long time that local anaesthetic affects the heart rate and blood pressure, however the investigators would like to describe exactly how, in much more detail.

ELIGIBILITY:
Inclusion Criteria:

* Any adult patient undergoing trans-sphenoidal pituitary surgery.

Exclusion Criteria:

* Under 16 years of age, pregnancy, uncontrolled hypertension, allergy to any local anaesthetic, patient refusal or revision pituitary surgery.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing trans-sphenoidal resection of a pituitary tumour.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2014-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure after administration of local anaesthesia | 5 minutes
  Changes in mean arterial pressure from baseline after infiltration of local anaesthetic.

SECONDARY OUTCOMES:
Change in heart rate after administration of local anaesthesia | 5 minutes
  Changes in mean arterial pressure from baseline after infiltration of local anaesthetic.
Change in cardiac output after administration of local anaesthesia | 5 minutes
  Changes in cardiac output from baseline after infiltration of local anaesthetic.
Change in systemic vascular resistance after administration of local anaesthesia | 5 minutes
  Changes in systemic vascular resistance from baseline after infiltration of local anaesthetic.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew D Wiles, FRCA FFICM, Study Chair — Sheffield Teaching Hospitals NHS Foundation Trust